CLINICAL TRIAL: NCT06962293
Title: Magnetic Anchor Guided - Endoscopic Submucosal Dissection (MAG-ESD) for Gastric and Colorectal Superficial Lesions - a Pilot Study
Brief Title: Magnetic Guided Counetrtraction During Endoscopic Submucosal Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2025.116
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Early Gastric Cancer; Colon Neoplasia
Keywords: endoscopic submucosal dissection; magnetic retractor
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAG-ESD assisted ESD (Experimental): Magnetic retractor assisted ESD performed
  Interventions: Device: MAG-ESD assisted ESD

INTERVENTIONS:
Device: MAG-ESD assisted ESD — Flexible magnetic traction device would be used to assist the ESD procedure. Real time adjustment of traction could be achieved by controlling the EPM position and orientation anytime during the procedure.

SUMMARY:
Endoscopic submucosal dissection (ESD) is a technique that allows curative treatment of early gastrointestinal neoplasia with organ preservation. However, it is a technically demanding procedure. Tissue traction plays a vital role in facilitating the visualization of the cutting line and the submucosal vessels, which usually only relies on the hood attached to the tip of the endoscope. However, when dealing with flat or large lesions, the absence of reliable traction in ESD contributes to its technical complexity and prolongs procedure duration. Various traction devices and techniques have been developed to provide tension for the dissection plane and optimal visibility during ESD. Most of these only provide static traction from a fixed angle, thus the effect of traction diminishes when the dissection continues.

In contrast to the aforementioned traction methods, magnetic traction offers the ability to externally manipulate an internal magnetic retractor, simplifying the internal workspace. The proposed magnetic retractor is composed of a detachable clip from an hemoclip is affixed to a magnetic element. By adjusting the position of the external magnetic source, the magnetic retractor automatically couples and aligns with it, enabling simultaneous dynamic directional control during the ongoing ESD operation. A novel robotic magnetic countertraction system was developed (MAG-ESD). The system consists of two sections: an external permanent magnetic source and the disposable magnetic retractor. The external permanent magnetic source is composed by a large external permanent magnet (EPM) which held by robot arm to externally control the locomotion of the magnetic retractor within patient. The disposable magnetic retractor is a consumable surgical instrument that modified from a commercial hemoclip, which has small magnets hangs on the clip legs. The design of the disposable magnetic retractor eliminates the need for endoscope withdrawal which can be inserted through the instrument channel from the handle during ESD operations, like other common instruments. In the current pilot study, the novel MAG-ESD counetrtraction system would be tested in 20 patients who undergo gastric and colonic ESD, with the aim of evaluating the system efficacy and safety.

DETAILED DESCRIPTION:
Gastrointestinal (GI) cancers accounted for 39.5 million new cases worldwide in 2020, representing 14.7% of the total new cases of cancer. These cancers also led to 18.8 million deaths, constituting 19% of the total deaths caused by cancer. Typically, endoscopic resection is recommended for early-stage tumors within the GI tract, with endoscopic submucosal dissection (ESD) often utilized for submucosal resection. Tissue traction plays a vital role in facilitating the visualization of the cutting line and the submucosal vessels. However, when dealing with flat or large lesions, the absence of reliable traction in ESD contributes to its technical complexity and prolongs procedure duration.

Various traction devices and techniques have been developed to provide tension for the dissection plane and optimal visibility during ESD. Examples include the "S-O clip" , "Ring thread", "Multiloop", "Double clip and rubber band" , etc. These methods typically involve the deployment of two or more clips to secure both the lesion site and the organ wall. The clips are constrained by springs or strings, allowing for control of the traction direction by deploying new clips to anchor the device at different locations. There is often a need to introduce a new clip through the instrument channel when adjusting the traction direction after the initial clips are anchored. Additional clips must be deployed to manipulate tissue traction, further complicates the internal working space, and inhibits the camera's peripheral vision. The traction achieved is not dynamic. Another drawback is that the traction force weakens during ongoing resection due to the elastic nature of the materials used, especially when the distance between the anchored clips decreases.

In contrast to the aforementioned traction methods, magnetic traction offers the ability to externally manipulate an internal magnetic retractor, simplifying the internal workspace. The proposed magnetic retractor is composed of a detachable clip from an hemoclip is affixed to a magnetic element. By adjusting the position of the external magnetic source, the magnetic retractor automatically couples and aligns with it, enabling simultaneous dynamic directional control during the ongoing ESD operation. Previous research has explored various designs of the magnetic element and external magnetic source. While many magnetic traction methods require withdrawing the endoscope to prepare the deployment of magnetic retractor.

Hence, a novel robotic magnetic countertraction system was developed (MAG-ESD). The system consists of two sections: an external permanent magnetic source and the disposable magnetic retractor. The external permanent magnetic source is composed by a large external permanent magnet (EPM) which held by robot arm to externally control the locomotion of the magnetic retractor within patient. The disposable magnetic retractor is a consumable surgical instrument that modified from a commercial hemoclip, which has small magnets hangs on the clip legs. The design of the disposable magnetic retractor eliminates the need for endoscope withdrawal which can be inserted through the instrument channel from the handle during ESD operations, like other common instruments. Additionally, a robot-assisted external permanent magnetic source can alleviate the workload of surgeons or assistants on controlling the movement of the EPM for the tissue traction inside patients. Robots assist in translating the heavy EPM with speed and low physical demand. An easily controlled magnetic retractor providing consistent traction force could significantly reduce the procedure time and enhance the process of ESD efficiency. The novel system has potential in reducing the procedure time and reducing the workload of endoscopists. The current pilot study aims to confirm the feasibility and safety of using this robotic magnetic countertraction system for MAG-ESD in patients with gastric and colorectal superficial lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient with superficial gastric or colorectal lesions, scheduled for endoscopic submucosal dissection (ESD).

Exclusion Criteria:

1. Patient who refused to participate
2. Other cases deemed by the examining physician as unsuitable for safe treatment

   The robotic magnetic countertraction system consist of a strong permanent magnet which always have a strong magnetic field in its surrounding. Therefore, we follow the MRI precautions for the strict safety measurement:
3. Patient who had a cardiac pacemaker.
4. Patient who had any metallic implant or device, such as drug pump, stent, etc.
5. Patient who has or had any metal fragments in eye or any other part of body, or had ever worked with metal.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-09 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | 1 day
  Successful en-bloc, without major intra-operative adverse event.

SECONDARY OUTCOMES:
Clinical success rate | 30 days
  pathological R0 resection, without major intra-operative and post-operative adverse event.
Total procedure time | 1 day
  Time taken from injection to completion of resection
MAG-ESD time | 1 day
  Time taken to apply the magnetic traction from introduction of magnetic retractor to the actual countertraction in effect
Lesion size | 1day
  Lesion size
Lesion location | 1 day
  Location of the lesion in the GI tract
NASA task load index | 1 day
  Endoscopist's NASA-TLX score for the procedure
Rate of all intraprocedural adverse event | 1 day
  Intra-procedural adverse event - total
Rate of intraprocedural adverse event - partial thickness muscle injury | 1 day
  Partial thickness muscle injury without full thickness perforation
Rate of intraprocedural adverse event - full thickness perforation | 1 day
  Full thickness perforation occurring intra-procedure
Rate of intra-procedural adverse event - haemorrhage | 1 day
  Major bleeding during procedure causing hemodynamic instability, or require blood transfusion, or causing haemoglobin drop >2g/dL
Rate of intraprocedural adverse event - other | 1 day
  Any other intraprocedural adverse event
Overall rate of Post-procedural adverse event | 30 days
  All post procedural adverse event
Rate of Post-procedural adverse event - delayed haemorrhage | 30 days
  Significant bleeding, with blood loss >2g/dL, or requiring blood transfusion, or causing hemodynamic instability, or requiring re intervention by endoscopy / surgery
Rate of post-procedural adverse event - delayed perforation | 30 days
  Delayed perforation occurring after completion of procedure
Rate of Post-procedural adverse event - post-ESD coagulation syndrome | 30 days
  Defined by presence of abdominal pain, and fever / leucocytosis after the procedure,
Rate of post-procedural adverse events - others | 30 days
  Any other adverse events after the procedure
Rate of complete resection (R0) | 30 days
  Resection specimen showing complete resection of the target lesion with negative histological horizontal and vertical margins
Rate of curative resection | 30 days
  Curative resection, defined based on Japanese gastroenterological endoscopy society (JGES) guidelines, depending on the tumor locations (Stomach and colorectal)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty of Medicine, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No